CLINICAL TRIAL: NCT03922399
Title: Outcome Evaluation for Burn Scar Therapy-laser and Surgery in Patients in Formosa Fun Coast Explosion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Principal Investigator, CHACHUN, CHEN, Plastic Surgeon, Shin Kong Wu Ho-Su Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20180606R
Record Dates: First submitted 2018-11-28; First posted 2019-04-22 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Patients With Major Burn Injury in Formosa FunCost Explosion
Keywords: burn scar; laser; ultrapulse
MeSH Terms: interventions — Laser Therapy

STUDY DESIGN:
Intervention Model Description: Patients with major burn scar, after lasers treatment for three years Evaluation tool: questionnaires, sonography, HRV
Masking Description: evaluating in different medical groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laser and Surgery in patients with major burn scars (Other): Evaluating patients with major burn scar after laser and surgical treatments Multiple-directions evaluation, including senior plastic resident, young resident, professional burn surgeons, senior nurse with burn scar, one non-medical patients(usually patients' family and friends)
  Interventions: Procedure: Laser and Surgery

INTERVENTIONS:
Procedure: Laser and Surgery — Laser and Surgery in patients with major burn scars Evaluating after three years treatment

SUMMARY:
Protocol title： Outcome evaluation for burn scar therapy-laser and surgery in patients in Formosa Fun Coast Explosion

Objectives： The goal of this study is to evaluate the effectiveness of both lasers and operations on patients with major burn scar(>20% TBSA).

DETAILED DESCRIPTION:
Background： There is no gold standard treatment for burn scar treatment, especially for those with major burn scar. In the Formosa Fun-Coast Dust Explosion in 2015, lots of patients with major burn scar suffer from severe pathologic burn scar syndromes. The gold of the study is to evaluate the efficacy of both lasers and operations on major burn scars treatment in the past two years.

Study Design： To take the assessment of scar into account, the investigators use both objectives and subjective methods to evaluate the scar condition. In addition to the scale of scar, the investigators also use both sonography and HRV system to evaluate the expressions of scar. All evaluated tools used are the same as those used in 20160201R and 20160202R. The investigators also used previous records to check the patient's scar condition before these treatments.

Hypothesis： After treatment, scar conditions should get better than before. However, the investigators need more scientific statistics to evaluate the improve rate.

Key words： Burn scar, burn scar syndromes. Scar laser treatment

ELIGIBILITY:
Inclusion Criteria:

1. >20% major burn scar, for 3 years
2. patients in Formosa FunCost Explosion
3. offering medical records, including laser and treatments
4. available for questionnaire evaluation and others' evaluation
5. those are willing to receive both sonography on scars and HRV evaluation

Exclusion Criteria:

1. those aren't willing to offer medical records
2. those aren't willing to fill questionnaire
3. those aren't willing to receive sonography on scars

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-01-27 (Actual); Study Completion 2019-03-08 (Actual)

PRIMARY OUTCOMES:
Patients objective questionnaire | Week 0
  Patients objective questionnaires is used to evaluate subjects' sensation and life quality, in which pain, itchiness and sleep are evaluated by Visual Analogue Scale (VAS), Burn Itchiness Scale and Sleep Assessment Scale, respectively.
Burn assessment by researchers | Week 0
  Burn scars are assessed using Vancouver scar scale by four plastic surgeons and a non-professional person.

SECONDARY OUTCOMES:
Scar evaluation by sonography (selective) | Week 0
  Burn scars in lower extremity are measured using 2-D problem sonography machine.
Autonomic nervous system analysis (selective) | Week 0
  Autonomic nervous system analysis is performed by heart-rate variability machine (HRV MACHINE).

CONTACTS AND LOCATIONS:
Locations (1):
- Shin Kong Wu Ho Su Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
lasers treatments, especially patients with major burn cases, are widely used. Therefore, we still consider the results after three years' treatments.